CLINICAL TRIAL: NCT05216120
Title: Efficacy and Safety of Pemigatinib in Subjects With Advanced Metastatic or Surgically Unresectable Adenosquamous Carcinoma of the Pancreas (ASCP) Who Have Progressed On Previous Therapy
Brief Title: Pemigatinib in Subjects With Adenosquamous Carcinoma of the Pancreas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: enrollment challenges
Sponsor: HonorHealth Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Incyte-54828-19-05
Record Dates: First submitted 2022-01-05; First posted 2022-01-31 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Pancreas Cancer
Keywords: pancreatic cancer; adenosquamous carcinoma of the pancreas; ASCP; phase II
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pemigatinib (Experimental): Participants will be provided with a bottle of pemigatinib tablets on Day 1 of each cycle (one cycle = 21 days). A bottle contains 4.5 mg X 42 tablets total. Each pemigatinib bottle is sufficient for one cycle. Resupply will be provided as necessary on Day 1 of each cycle.
  Interventions: Drug: Pemigatinib 4.5 MG

INTERVENTIONS:
Drug: Pemigatinib 4.5 MG — Pemigatinib 4.5 mg tablets taken 3 times per day [daily dose of 13.5 mg (3 tablets)] for 14 consecutive days followed by 7 days off medication in 21-day cycles
  Doses will be self-administered at home. Participants will be instructed to take study medication at the same time each day, with or without food.
  Other Names: Pemazyre

SUMMARY:
The purpose of this research is to determine the benefit of pemigatinib in patients with advanced metastatic or surgically unresectable adenosquamous carcinoma of the pancreas who have progressed on previous therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age; male or female
* Capable of providing informed consent and complying with trial procedures.
* Histologically or cytologically confirmed adenosquamous carcinoma of the pancreas (ASCP)
* Metastatic or unresectable ASCP patients who have progressed on at least one line of therapy
* FGFR gene fusion, mutation, or rearrangement as determined by standard CLIA-certified FDA-approved genomic panel (e.g. Ashion, Caris, FoundationOne etc.).
* Radiographically measurable or evaluable disease according to RECIST 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Life expectancy ≥ 12 weeks.
* Females of child-bearing potential (defined as a sexually mature woman who (1) has not undergone hysterectomy [the surgical removal of the uterus] or bilateral oophorectomy [the surgical removal of both ovaries] or (2) has not been naturally postmenopausal for at least 24 consecutive months [i.e., has had menses at any time during the preceding 24 consecutive months]) must:

  1. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis), or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting study treatment (including dose interruptions), and while on study treatment and for 1 week following discontinuation from study treatment ;and,
  2. Have a negative serum pregnancy test (β -hCG) result at screening and agree to ongoing pregnancy testing during the course of the study, and at the end of study participation. This applies even if the subject practices true abstinence* from heterosexual contact.
* Male subjects must practice true abstinence* or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for 1 week following discontinuation from study treatment, even if he has undergone a successful vasectomy.

Exclusion Criteria:

* Patients that have received prior treatment with a selective FGFR inhibitor
* History of and/or current evidence of ectopic mineralization/calcification, including but not limited to soft tissue, kidneys, intestine, myocardia, or lung, excepting calcified lymph nodes and asymptomatic arterial or cartilage/tendon calcifications.
* Current evidence of clinically significant corneal or retinal disorder confirmed by ophthalmologic examination.
* Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives, whichever is shorter, before the first dose of study drug. Topical ketoconazole will be allowed.
* Exposure to any therapeutic or investigational agent(s) within 3 weeks prior to initiation of study treatment.
* Major surgery within 4 weeks prior to initiation of study treatment.
* Any condition in the opinion of the principal investigator that might interfere with the patient's participation in the study or in the evaluation of the study results.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate of pemigatinib | Initiation of study treatment up to 12 cycles (each cycle is 21 days)
  Overall response rate of pemigatinib in patients with advanced metastatic or surgically unresectable ASCP who have progressed on previous therapy

SECONDARY OUTCOMES:
Progression free survival (PFS) | Initiation of study treatment up to study completion, up to 2 years
  To determine progression free survival (PFS)
Overall survival (OS) | Initiation of study treatment up to study completion, up to 2 years
  To determine overall survival (OS)
Number of participants with treatment-related adverse events as assessed by CTCAE V4.0 | Initiation of study treatment up to 12 cycles (each cycle is 21 days)
  To determine the overall safety (medical risk to the subject) and tolerability (the degree to which adverse effects can be tolerated by the subject) of pemigatinib in patients with advanced metastatic or surgically unresectable ASCP who have progressed on previous therapy

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Borazanci, MD, Principal Investigator — HonorHealth Research Institute
Locations (1):
- HonorHealth Research Institute, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No